CLINICAL TRIAL: NCT00000878
Title: A Phase I/II, Open-Label Study to Evaluate the Safety, Tolerance and Pharmacokinetics of Stavudine (d4T) in Combination With Lamivudine (3TC) in HIV-Infected Pregnant Women and Their Infants
Brief Title: A Study to Evaluate the Safety and Tolerance of Stavudine (d4T) in Combination With Lamivudine (3TC) in HIV-Positive Pregnant Women and Their Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 332; 11304 (Registry Identifier: DAIDS ES); PACTG 332
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Pregnancy Complications, Infectious; Drug Therapy, Combination; Stavudine; Lamivudine; Disease Transmission, Vertical; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious | interventions — Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to evaluate the safety and tolerance of 2 anti-HIV drugs, d4T and 3TC, given in combination to HIV-positive pregnant women and their infants.

Most HIV-positive pregnant women usually take the anti-HIV drug zidovudine (ZDV) to treat HIV and reduce the chances of giving HIV to their babies. It recently has been shown that a combination of drugs may be more effective than ZDV alone. This study tests the effectiveness of combinations of ZDV, d4T, and 3TC.

DETAILED DESCRIPTION:
New antiretroviral agents or combinations are sought that are as efficacious as ZDV and that would be effective in reducing the rate of vertical transmission of HIV in women who have been long-term recipients of ZDV. d4T is a good candidate drug. It is a thymidine nucleoside analogue that inhibits replication of HIV at concentrations similar to those of ZDV which have anti-HIV activity. The demonstrated safety profile of d4T, the ease of administration, and, most importantly, preliminary efficacy data, especially in combination with 3TC, make this an excellent candidate combination for a Phase I perinatal trial.

Two cohorts of women and infants are enrolled in this study. The first five mother/infant pairs enrolled comprise Group I. Mothers enrolled in this group must allow their infants to receive ZDV. Eight mother/infant pairs are then enrolled in Group II; Group II infants are allocated into two groups: those whose mothers allow the administration of ZDV (Group IIA) and those whose mothers do not (Group IIB).

Group I:

Women:

Beginning at a minimum of 14 weeks gestation:

1. Oral d4T until the start of active labor.
2. Oral 3TC.

At the start of active labor (defined as regular uterine contractions resulting in cervical dilation [3-4 cm] and effacement [50-60%]) and during delivery:

1. d4T administered IV as a loading dose followed by a continuous infusion until the umbilical cord is clamped.
2. Oral 3TC if patient's previous dose of 3TC was administered at least 0.5h prior to onset of labor and additional dose of 3TC is administered and the time until next dose is scheduled accordingly.

Infants:

1. d4T as a single oral dose on Day 6 (+/- 2 days) and on Day 42 (this dose can be given between Days 35 and 42, inclusive).
2. Oral ZDV (or IV if unable to take oral dosing) for 6 weeks, beginning a maximum of 12 hours after birth.
3. 3TC for 6 weeks, beginning a maximum of 12 hours after birth.

Group II:

Women:

Beginning at a minimum of 14 weeks gestation:

1. Oral d4T until the umbilical cord is clamped.
2. Oral 3TC.

At the start of active labor and through delivery:

Oral d4T and 3TC as above. If the last doses of d4T and 3TC were given at least 0.5 hours prior to onset of active labor, an additional dose of d4T and 3TC is given and repeated every 12 hours.

Infant Group IIA:

1. d4T as a single oral dose on Day 6 (+/- 2 days) and on Day 42 (this dose can be given between Days 35 and 42, inclusive).
2. Oral ZDV (or IV if unable to tolerate oral dosing) for 6 weeks, beginning a maximum of 12 hours after birth.
3. 3TC for 6 weeks, beginning a maximum of 12 hours after birth.

Infant Group IIB:

Beginning a maximum of 12 hours after birth:

1. d4T for 6 weeks.
2. 3TC for 6 weeks. [AS PER AMENDMENT 9/15/97: If tolerated, infants continue on protocol treatment to 6 weeks of age. At 6 weeks, infants should receive standard care, including PCP prophylaxis, from an HIV specialist/pediatrician. HIV-infected infants are offered ACTG trial enrollment or open-label treatment based on best clinical judgment of their physician.] [AS PER AMENDMENT 2/19/99: Patients who prematurely discontinue study treatment should continue to be followed on study for the duration of the study.]

ELIGIBILITY:
Inclusion Criteria

Women may be eligible for this study if they:

* Are HIV-positive.
* Are at least 13 years old (need consent of parent or guardian if under 18).
* Are unable to or refuse to take ZDV or the woman's doctor says that she should take d4T.
* Are 14 to 34 weeks pregnant.

Exclusion Criteria

Women will not be eligible for this study if they:

* Have a history of peripheral neuropathy.
* Have an active opportunistic infection and/or serious bacterial infection within 14 days of study entry.
* Have severe diarrhea.
* Are allergic to d4T or 3TC.
* Use illicit drugs or abuse alcohol.
* Are taking anti-HIV drugs other than study medications.
* Are planning to breast-feed.
* Are having a problem pregnancy (baby is not developing correctly or will not survive birth) or have had pregnancy complications in the past.
* Babies will not be eligible for this study if they:
* Are unable to take medications by mouth for more than 72 hours.
* Have severe birth defects or other life-threatening conditions.
* Are underweight (less than 2 kg).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26
Dates: Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Wade, Study Chair; Sandra Burchett, Study Chair; Salih Yasin, Study Chair; Jash Unadkat, Study Chair
Locations (20):
- United States (18):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Children's Hosp of Boston, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Temple Univ School of Medicine, Philadelphia, Pennsylvania
  - Regional Med Ctr at Memphis, Memphis, Tennessee
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (2):
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan